CLINICAL TRIAL: NCT05876949
Title: A Randomized, Double-blind, Parallel Design, Single Dose, 2-arm Study Comparing the Pharmacokinetic, Safety and Immunogenicity Profiles of AVT03 and US-Xgeva® in Healthy Male Subjects
Brief Title: AVT03 With Xgeva in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alvotech Swiss AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: AVT03-GL-P03
Record Dates: First submitted 2023-05-17; First posted 2023-05-26 (Actual); Results first posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-04

CONDITIONS: This is a Phase I Study Conducted in Healthy Volunteers
Keywords: Denosumab; Healthy Volunteers
MeSH Terms: interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Experimental Arm AVT03 120mg (Experimental): AVT03 is the proposed biosimilar for Xgeva (denosumab). Subjects in this arm will receive a single 120mg dose of AVT03 as a subcutaneous injection
  Interventions: Biological: AVT03
- Active Comparator Xgeva 120mg (Active Comparator): Xgeva (denosumab) is the proposed active comparator for AVT03. Subjects in this arm will receive a single 120mg dose of Xgeva (denosumab) as a subcutaneous injection
  Interventions: Biological: Denosumab

INTERVENTIONS:
Biological: AVT03 — AVT03 will be given as 1 time subcutaneous injection
  Other Names: AVT03 proposed Biosimilar to Denosumab
  Arms: Experimental Arm AVT03 120mg
Biological: Denosumab — Xgeva (denosumab) will be given as 1 time subcutaneous injection
  Other Names: Xgeva
  Arms: Active Comparator Xgeva 120mg

SUMMARY:
This study has been designed as a randomized, double-blind, parallel-group study and in healthy adult male subjects of age 28 years to 55 years old. The study will assess the PK, safety and tolerability of AVT03 compared to US-Xgeva when administered as a single 120 mg SC dose

DETAILED DESCRIPTION:
The study will consist of screening period, a 196 day (28 weeks) treatment and assessment period, and an End of Study (EOS) visit on week 32 on Day 196. Subjects will undertake a screening visit between Day -28 and Day -1 to determine their eligibility for the study. Subjects who meet the eligibility criteria will be admitted to the study site on the day prior to dosing (Day -1), during which their continued eligibility will be assessed up to Day 1 prior to dosing. On Day 1, eligible subjects will be randomized and will receive a single dose of 120mg AVT03 or 120mg Xgeva as subcutaneous injection.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
2. Male subjects who are 28 to 55 years old, inclusive, at the time of signing the ICF.
3. Have a body weight of 50.0 to 90.0 kg (inclusive) and body mass index of 17.0 to 32 kg/m2 at Screening and Day -1.

Exclusion Criteria:

1. Evidence of clinically relevant pathology, especially prior diagnosis of bone disease, or any uncontrolled condition that will affect bone metabolism such as, but not limited to: osteoporosis, osteogenesis imperfecta, hyperparathyroidism,, non-controlled hyperthyroidism osteomalacia, rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, current flare-up of osteoarthritis and/or gout, active malignancy, renal disease, Paget's disease of the bone, malabsorption syndrome.
2. Have osteonecrosis of the jaw (ONJ) or risk factors for ONJ such as invasive dental procedures (e.g., tooth extraction, dental implants, oral surgery) or intend to undergo such procedures during the study period, poor oral hygiene, periodontal, and/or pre-existing dental disease.
3. Have bone fractures, presence of active healing fractures, or recent bone fracture
4. Abnormal serum calcium.
5. Known vitamin D deficiency.

Ages: 28 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 208 (Actual)
Dates: Start 2023-07-21 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Felicitas Bullo, Study Director — Alvotech Swiss AG
Locations (3):
- Biokinetica, Józefów, Poland
- Farmovs, Bloemfontein, South Africa
- Richmond Pharmacology, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tomaszewska-Kiecana M, Bullo F, Jaskiewicz L, Stamatakos S, Otto H, Rai M, Sattar A, Leutz S, Berti F. A randomized, double-blind, single dose, parallel group, 2-arm study assessing the pharmacokinetic similarity, safety, tolerability, and immunogenicity profiles of biosimilar candidate AVT03 (70 mg/mL) in healthy male adults. Expert Opin Investig Drugs. 2025 Jun;34(6):539-546. doi: 10.1080/13543784.2025.2505469. Epub 2025 May 16. PMID 40357869

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental Arm AVT03 120mg: AVT03 is the proposed biosimilar for Xgeva (denosumab). Subjects in this arm received a single 120mg dose of AVT03 as a subcutaneous injection
  AVT03 was given as 1 time subcutaneous injection
- Active Comparator Xgeva 120mg: Xgeva (denosumab) is the proposed active comparator for AVT03. Subjects in this arm received a single 120mg dose of Xgeva (denosumab) as a subcutaneous injection
  Denosumab: Xgeva (denosumab) was given as 1 time subcutaneous injection
Period: Overall Study
Arm/Group | Experimental Arm AVT03 120mg | Active Comparator Xgeva 120mg
Started | 104 | 104
Completed | 103 | 98
Not Completed | 1 | 6
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Physician Decision | 0 | 2
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants were healthy males aged 28 to 55 years.
Groups:
- Experimental Arm AVT03 120mg: AVT03 is the proposed biosimilar for Xgeva (denosumab). Subjects in this arm received a single 120mg dose of AVT03 as a subcutaneous injection
  AVT03: AVT03 was given as 1 time subcutaneous injection
- Active Comparator Xgeva 120mg: Xgeva (denosumab) is the active comparator for AVT03. Subjects in this arm received a single 120mg dose of Xgeva (denosumab) as a subcutaneous injection
  Denosumab: Xgeva (denosumab) was given as 1 time subcutaneous injection
- Total: Total of all reporting groups
Arm/Group | Experimental Arm AVT03 120mg | Active Comparator Xgeva 120mg | Total
Number analyzed (Participants) | 104 | 104 | 208
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.5 (6.72) | 38.1 (7.08) | 37.3 (6.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 104 | 104 | 208
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian (Japanese) | 12 | 12 | 24
  Black or African American | 28 | 24 | 52
  Caucasian/White | 64 | 68 | 132

OUTCOME MEASURES:

1. Primary Outcome: Co-primary PK Endpoint Cmax: Maximum Serum Concentration
Description: Samples will be collected for measurement
Time Frame: Day 1 (pre-dose, 8h and 12h post-dose), Day 2 to Day 13 (daily), Day 15, Day 18, Day 22, Day 25, Day 29, Day 43, Day 57, Day 71, Day 85, Day 99, Day 112, Day 126, Day 141, Day 162 and Day 196 (week 28) / End of study
Population: A total of 4 participants were excluded from the PK population analyses set (1 participant in the AVT03 group and 3 participants in the Xgeva group) due to limited duration of PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Experimental Arm AVT03 120mg | Active Comparator Xgeva 120mg
Number analyzed (Participants) | 103 | 101
ng/mL | 12761.4 (34) | 12259.8 (32)

2. Primary Outcome: Co-primary PK endpoint_AUC0-t: Area Under the Serum Concentration-time Curve up to Time t, Where t is the Last Time Point With a Concentration Above the Lower Limit of Quantitation
Description: Samples will be collected for measurement
Time Frame: as for outcome 1
Population: A total of 4 participants were excluded from the PK population analyses set (1 participant in the AVT03 group and 3 participants in the Xgeva group) due to limited duration of PK data.[
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: ng·h/mL
Arm/Group | Experimental Arm AVT03 120mg | Active Comparator Xgeva 120mg
Number analyzed (Participants) | 103 | 101
ng·h/mL | 15501387.9 (27) | 14366056.2 (29)

3. Secondary Outcome: PK_ AUC0-inf: Comprised of AUC0-t and AUC Extrapolated From Time t to Time Infinity.
Description: Samples will be collected for measurement
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng·h/mL
Arm/Group | Experimental Arm AVT03 120mg | Active Comparator Xgeva 120mg
Number analyzed (Participants) | 103 | 101
ng·h/mL | 15559245.8 (28) | 14555779.3 (29)

4. Secondary Outcome: Safety Incidence, Nature and Severity of Adverse Events.
Time Frame: Day 1(week 1) to Day 196 (week 28)]
Measure: Number; unit: participants
Arm/Group | Experimental Arm AVT03 120mg | Active Comparator Xgeva 120mg
Number analyzed (Participants) | 104 | 104
participants
  Any TEAE | 66 | 67
  TESAEs | 1 | 3

5. Secondary Outcome: Immunogenicity Presence of ADAs and Presence of nAbs Against AVT03 and Xgeva
Description: Samples will be collected for measurement
Time Frame: Day 1, Day 8, Day 15, Day 29, Day 57, Day 71, Day 112, Day 141, Day 196/EoS
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Arm AVT03 120mg | Active Comparator Xgeva 120mg
Number analyzed (Participants) | 104 | 104
Participants
  Binding (ADA) | 104 | 102
  Neutralizing Antibodies | 41 | 43

ADVERSE EVENTS:
Time Frame: All AEs/SAEs were recorded from the time of signing the ICF until the end of the subject's participation in the study, up to 32 weeks.
Arm/Group | Experimental Arm AVT03 120mg | Active Comparator Xgeva 120mg
All-Cause Mortality (participants affected / at risk) | 0/104 | 1/104
Serious Adverse Events (participants affected / at risk) | 1/104 | 3/104
Other Adverse Events (participants affected / at risk) | 66/104 | 67/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Arm AVT03 120mg (N=104) | Active Comparator Xgeva 120mg (N=104)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Small bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Alcohol use disorder (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Arm AVT03 120mg (N=104) | Active Comparator Xgeva 120mg (N=104)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 5 (7) | 1 (2)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 2 (2)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Chalazion (Eye disorders) | 0 (0) | 1 (2)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Tongue ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 2 (2)
Application site rash (General disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Hyperthermia (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 3 (4) | 2 (3)
Injection site erythema (General disorders) | 2 (2) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 3 (3) | 4 (5)
Injection site swelling (General disorders) | 1 (1) | 0 (0)
Swelling face (General disorders) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Body tinea (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2)
COVID-19 (Infections and infestations) | 1 (1) | 4 (4)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Enterobiasis (Infections and infestations) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 2 (2) | 4 (4)
Genital herpes (Infections and infestations) | 0 (0) | 1 (2)
Gonococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Groin abscess (Infections and infestations) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 5 (5) | 6 (6)
Nasopharyngitis (Infections and infestations) | 11 (12) | 11 (13)
Oral herpes (Infections and infestations) | 2 (2) | 3 (3)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pulpitis dental (Infections and infestations) | 1 (1) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 11 (11) | 10 (10)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Viraemia (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injury corneal (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Penis injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 8 (8) | 5 (7)
Blood potassium increased (Investigations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 5 (5) | 2 (4)
Blood triglycerides increased (Investigations) | 1 (1) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 10 (12) | 7 (8)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Tension headache (Nervous system disorders) | 0 (0) | 1 (2)
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Bleeding varicose vein (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-11): https://cdn.clinicaltrials.gov/large-docs/49/NCT05876949/Prot_SAP_000.pdf